CLINICAL TRIAL: NCT05734495
Title: A Phase II Study Evaluating Venetoclax and Pirtobrutinib in Previously Treated Waldenström Macroglobulinemia
Brief Title: Pirtobrutinib and Venetoclax in Waldenström Macroglobulinemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jorge J. Castillo, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-611
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom Macroglobulinemia; Lymphoplasmacytic lymphoma
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — pirtobrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PIRTOBRUTINIB + VENETOCLAX (Experimental): Participants will receive:
  * Standard of care bone marrow aspirate & biopsy within 90 days of Cycle 1 Day 1.
  * Computed Tomography (CT) scan of chest, pelvis & abdomen within 90 days of Cycle 1 Day 1.
  * Electrocardiogram at screening.
  * Cycle 1
    * Electrocardiogram.
    * Day 1-28: Predetermined dose of Pirtobrutinib 1x daily.
  * Cycle 2
    -Day 1-28: Predetermined dose Pirtobrutinib & Venetoclax 1x daily. Tumor lysis syndrome (TLS) prophylaxis, predetermined dose Allopurinol at least 72 hrs prior to 1st administration of Venetoclax and dose escalation at Day 8 & Day 15.
  * Cycles 3-24
    * Day 1-28: Predetermined dose of Pirtobrutinib & Venetoclax 1x daily.
    * Electrocardiogram: Cycles 3, 6, 9,12,15,18,21,24
    * CT scan of chest, pelvis & abdomen: Cycles 7, 13, End of Treatment if extramedullary disease at baseline unresolved in previous CT scan
    * Standard of care bone marrow aspirate and biopsy: Cycles 7, 13, End of Treatment
  * Follow up every 12 wks for 4 yrs.
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Pirtobrutinib — Noncovalent Bruton Tyrosine Kinase (BTK) inhibitor, tablet taken orally.
  Other Names: LY3527727, LOXO-305
Drug: Venetoclax — Small-molecule B-cell lymphoma-2 (Bcl-2) family inhibitor, tablet taken orally.
  Other Names: ABT-199, A-1195425.0, GDC-0199, RO5537382, Venclexta, and Venclyxto.

SUMMARY:
This study is being done to examine the safety and effectiveness of pirtobrutinib combined with venetoclax as a possible treatment for participants with Waldenström Macroglobulinemia (WM).

The names of the study drugs involved in this study are:

* Pirtobrutinib (a Noncovalent Bruton Tyrosine Kinase (BTK) inhibitor)
* Venetoclax (a BCL2 inhibitor)

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase II study to evaluate the safety and efficacy of venetoclax combined with pirtobrutinib (VEN-P) in participants with symptomatic Waldenström Macroglobulinemia (WM) with previously treated disease. Pirtobrutinib blocks a type of protein called Bruton Tyrosine Kinase (BTK) that helps cells live and grow. Venetoclax blocks BCL-2, a protein essential for WM cells' survival.

The U.S. Food and Drug Administration (FDA) has not approved pirtobrutinib for Waldenström Macroglobulinemia (WM), but it has been approved for other uses.

The FDA has not approved venetoclax for Waldenström Macroglobulinemia (WM), but it has been approved for other uses.

The FDA has not approved the combination of pirtobrutinib and venetoclax as a treatment for any disease.

Study procedures include screening for eligibility, treatment visits, CT scans, blood tests, and bone marrow aspirates and biopsies.

Participants will receive study treatment for up to 2 years and will be followed for up to 4 years or until they start a new therapy.

It is expected that about 42 people will take part in this research study.

Eli Lilly supports this research study by providing study drug pirtobrutinib and funding.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate. Screening evaluations including consent, physical exam, and laboratory assessments will be done within 30 days prior to Cycle 1 Day 1. Bone marrow biopsy & aspirate, and CT C/A/P will be done within 90 days prior to Cycle 1 Day 1.

* Clinicopathological diagnosis of Waldenström Macroglobulinemia, including MYD88 Wild-Type.
* At least 1 prior line of treatment.

  * Prior covalent BTK inhibitor is allowed even if prior progression documented on this agent.
  * Prior venetoclax is allowed unless participant had documented progression while on this agent.
* Symptomatic disease meeting criteria for treatment using consensus panel criteria from the Second International Workshop on WM. At least one of the following:

  --Constitutional Symptoms
  * Recurrent fever
  * Night sweats
  * Fatigue
  * Weight loss
  * Progressive or symptomatic lymphadenopathy or splenomegaly
  * Hemoglobin ≤ 10 g/dL
  * Platelet count ≤ 100 k/uL
  * Hyperviscosity syndrome
  * Symptomatic peripheral neuropathy
  * Systemic amyloidosis
  * Renal Insufficiency
  * Symptomatic cryoglobulinemia
* Age 18 years or older
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum serum IgM level of > 2 times the upper limit normal.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Women of childbearing potential: Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 6 months after discontinuation from the study. FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential (FCBP) even if they have had a successful vasectomy 1) while participating in the study; and 2) for at least 6 months after discontinuation from the study.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥750/ uL the patient may enroll below this threshold if there is documented bone marrow involvement considered to impair hematopoiesis
  * Platelets ≥50,000/ uL not requiring transfusion support; the patient may enroll below this threshold if there is documented bone marrow involvement considered to impair hematopoiesis
  * Hemoglobin ≥ 8 g/dL not requiring transfusion support or growth factors; the patient may enroll below this threshold if there is documented bone marrow involvement considered to impair hematopoiesis or hemolysis
  * Total bilirubin ≤ 1.5 X ULN, or ≤3 x ULN with documented liver involvement, hemolysis, or Gilbert's Disease
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal, or ≤5 X ULN with documented liver involvement
  * Creatinine clearance ≥ 30 ml/min using Cockcroft/Gault formula
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior exposure to non-covalent BTK inhibitors
* Participants who experienced a major bleeding event or grade > 3 arrhythmia on prior treatment with a BTK inhibitor. NOTE: Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2g per deciliter; or bleeding in a critical area or organ (e.g. retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome).
* Participants who are receiving any other investigational agents.
* Female participants who are pregnant, breastfeeding, or planning to become pregnant or breastfeed while enrolled in this study or within 6 months of last dose of study drug.
* Participants with known CNS lymphoma.
* Participants with known history of Human Immunodeficiency Virus (HIV) and known active cytomegalovirus (CMV) infection.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below:

  * Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (antiHBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation before enrollment. Patients who are hepatitis B PCR positive will be excluded.
  * Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before enrollment. Patients who are hepatitis C RNA positive will be excluded.
* Concurrent administration of warfarin.
* Concurrent administration of moderate or strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers and/or strong p-glycoprotein (P-gp) inhibitors
* Concurrent systemic immunosuppressant therapy. System steroids at doses <20mg prednisone per day are permitted.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Active uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the Investigator and the Sponsor makes it undesirable for the patient to participate in the trial. Screening for chronic conditions is not required.
* Major surgery within 4 weeks of first dose of study drug.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Participants with known history of alcohol or drug abuse.
* Participants with inability to swallow pills and inability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of the study participation
* Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) where new therapy introduced or concomitant therapy escalated within the 4 weeks prior to study enrollment is required to maintain adequate blood counts.
* Prolongation of the QT interval corrected for heart rate (QTcF) > 470 msec on at least 2/3 consecutive electrocardiograms (ECGs), and mean QTcF > 470 msec on all 3 ECGs, during Screening. QTcF is calculated using Fridericia's Formula (QTcF): QTcF=QT/(RR0.33).

  * Correction of suspected drug-induced QTcF prolongation can be attempted at the Investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
  * Correction for underlying bundle branch block (BBB) allowed. Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
* Significant cardiovascular disease defined as:

  * Unstable angina, or
  * History of myocardial infarction within 6 months prior to planned start of pirtobrutinib, or
  * Previously documented left ventricular ejection fraction (LVEF) by any method of ≤ 45% in the 12 months prior to planned start of pirtobrutinib; assessment of LVEF via echocardiogram or multigated acquisition (MUGA) scan during Screening should be performed in selected patients as medically indicated, or
  * Any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or
  * Uncontrolled or symptomatic arrhythmias
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, EKG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the patient; alter the absorption, distribution, metabolism or excretion of the study drug; or impair the assessment of study results
* Participants with a known hypersensitivity to any of the excipients of pirtobrutinib or venetoclax
* Participants with a history of non-compliance to medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2029-01-25 (Estimated); Study Completion 2033-01-25 (Estimated)

PRIMARY OUTCOMES:
Very Good Partial Response (VGPR) or Better Response Rate | up to 2 years
  VGPR or better response rate is defined as proportion of participants experienced VGPR or complete response (CR) based on modified 6th International Workshop on WM [IWWM] criteria (NCCN 2014).

SECONDARY OUTCOMES:
Best Response | up to 2 years
  Best response on treatment including complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), stable disease (SD) and progressive disease (PD) per Modified 6th IWWM (NCCN 2014) response criteria.
Median Progression-Free Survival (PFS) | up to 4 years
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last disease assessment.
Median Time to Next Treatment (TTNT) | Up to 6 years
  TTNT estimated using the Kaplan Meier method is defined as the duration of time from the first dose of pirtobrutinib until the time of initiation of new therapy, or censored at the date of last contact if no further new therapy initiated.
Median Duration of Response (DOR) | up to 4 years
  DOR estimated using the Kaplan Meier method, is defined as the duration of time from the day the criteria are met for response (at least a minor response) to the date that Progressive Disease (PD) or death are objectively documented. Response and PD defined protocol section 11.1.2 - Modified 6th IWWM (NCCN 2014) criteria. If a participant is still responding, then the participant's data will be censored at the last study visit at which a tumor assessment was performed.
Median Overall Survival (OS) | Up to 6 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Number of Participants Present MYD88 Mutation Status | Baseline to 4 years post-treatment
  MYD88 mutation status determined based on allele-specific polymerase-chain-reaction (PCR) assay.
Number of Participants Present CXCR4 Mutation Status | Baseline to 4 years post-treatment
  CXCR4 mutation status determined based on Sanger sequencing.
Number of Participants Present BTK Mutation Status | Baseline to 4 years post-treatment
  BTK mutation status determined based on allele-specific polymerase-chain-reaction (PCR) assay.
Number of Participants Present BCL2 Mutation Status | Baseline to 4 years post-treatment
  BCL2 mutation status determined based on allele-specific polymerase-chain-reaction (PCR) assay.
Quality of Life (QOL) | Baseline to up to 6 years from treatment initiation
  Changes in QOL score will be assessed using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30. The QLQ-C30 summary score is calculated as the mean of the combined 13 QLQ-C30 scale and Item scores, with a higher score indicating a better QOL.
Grade 3-5 Treatment-related Toxicity Rate | up to 25 months
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAE v5 as reported on case report forms will be counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Castillo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconness Medical, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu